CLINICAL TRIAL: NCT06308627
Title: A One-year Trajectory of Depression Status Changes in Older Adults With Mild Cognitive Impairment and Subthreshold Depression: a Longitudinal Cohort Study
Brief Title: A One-year Trajectory of Depression Status Changes in Older Adults With MCI and SD: a Longitudinal Cohort Study
Status: Completed | Type: Observational
Sponsor: Fujian Medical University (Other)
Responsible Party: Principal Investigator, Dan Ting Chen, Principal Investigator, Fujian Medical University
Other Study IDs: K2022-03-074
Record Dates: First submitted 2024-03-04; First posted 2024-03-13 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Mild Cognitive Impairment; Subthreshold Depression; Older Adults
Keywords: Mild Cognitive Impairment; Subthreshold Depression; Older adults
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to investigate the one-year trajectory of changes in depression status in older adults with mild cognitive impairment and subthreshold depression, and to explore relevant risk factors for predicting changes in depression status. This one-year prospective longitudinal follow-up study involved 400 (expected) subjects who met the diagnostic criteria for mild cognitive impairment combined with subthreshold depression in older adults, and their depressive status was assessed using the Geriatric Depression Scale (GDS). Follow up monitoring of depression status at 6 and 12 months. Obtain factors related to changes in depressive status (such as age, gender, education level, cognitive function, anxiety level, sleep status, social support, psychological resilience, social network, etc.). By studying the longitudinal trajectory of depression status in elderly patients with mild cognitive impairment and subthreshold depression, a multi state Markov model with time and state discreteness is constructed, namely: State 1 (normal); State 2 (subthreshold depression); State 3 (mild depression); State 4 (moderate depression); State 5 (severe depression). Deeply explore and analyze the impact of certain factors and indicators on the transition between states, and estimate the probability of transition between states.

ELIGIBILITY:
Inclusion Criteria:

1. Age: ≥ 60 years old
2. Meets the diagnostic criteria for mild cognitive impairment and subthreshold depression
3. Having basic comprehension and verbal expression skills
4. Voluntarily participate in this study and sign an informed consent form.

Exclusion Criteria:

1. Diagnosed as depression patients, including patients with organic mental disorders and patients with a history of depression related mental disorders
2. Cognitive impairment caused by other diseases (such as neurological and psychiatric disorders, metabolic disorders, poisoning, infections, etc.)
3. Severe heart, liver, and kidney diseases
4. Serious chronic diseases and complications, such as congestive heart failure, hypertension, diabetes and other diseases with serious complications

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Select elderly patients with mild cognitive impairment and subthreshold depression who meet the inclusion and exclusion criteria from multiple elderly care institutions, a tertiary hospital in Fuzhou, and communities in Fujian Province as the research subjects.
Sampling Method: Non-Probability Sample
Enrollment: 466 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Depressive state | 2023.6.1-2024.7.1
  The Geriatric Depression Scale (GDS-15) is used to investigate the psychological feelings of patients in the past week. Result evaluation criteria: The total score range is 0-15 points, with higher scores indicating more severe depression. 1-5 points are subthreshold depression, 6-7 points are mild depression, 8-11 points are moderate depression, and 12-15 points are severe depression.

SECONDARY OUTCOMES:
General information of patients | 2023.6.1-2024.7.1
  Using a self-made general information scale, such as age, gender, education level, and other basic personal information
Cognitive | 2023.6.1-2024.7.1
  Montreal Cognitive Assessment (MoCA) is an assessment tool used for rapid screening of mild cognitive impairment. The total score is 30 points, and the higher the score, the better the cognitive function of the research subject. Literacy group ≤ 13 points, primary school group ≤ 19 points, and middle school and above group ≤ 24 points can be judged as cognitive impairment.
Activity of Daily Living | 2023.6.1-2024.7.1
  The Activities of Daily Living (ADL) scale adopts a Liket four level rating. The evaluation results can be analyzed based on total score, dimension score, and individual score. A total score of 20 is considered completely normal, while a score above 20 indicates varying degrees of functional decline. A score of 1 for each item indicates normal functionality, while a score of 2-4 indicates decreased functionality.
Anxiety | 2023.6.1-2024.7.1
  The Self Rating Anxiety Scale (SAS) has a total of 20 items, of which 5, 9, 13, 17, and 19 items are scored in reverse. The scale adopts a 1-4 level scoring method (1 point for no or very little time; 2 points for a small portion of time; 3 points for a considerable amount of time; 4 points for the vast majority or all of time). Individuals fill in the scale based on their own situation in the most recent week, multiply the calculated total score by 1.25, take an integer as the standard score, and use it as a statistical indicator. The higher the standard score, the more severe the anxiety level of the individual.
Social Function | 2023.6.1-2024.7.1
  The Social Support Rating Scale (SSRS) includes three dimensions: objective support, subjective support, and support utilization, with a total of 10 items: 1 point (none) to 4 points (full support). The higher the score in each dimension, the more support received.
Social Function | 2023.6.1-2024.7.1
  The Lubben Social Network Scale (LSNS-6) is used to measure the structural characteristics of individual family and friend networks, as well as the supporting functions played by the network, in order to reflect the social network level of the respondents. It consists of two parts: the home network and the friend network, each with three items, totaling six items. Each entry has 5 options, with a score of 0-5 points and a total score of 0-30 points. The higher the score, the higher the level of social network, and<12 points indicates insufficient social network.
Sleep Quality | 2023.6.1-2024.7.1
  The Pittsburgh Sleep Quality Index (PSQI) has a total of 19 items, divided into 7 components: subjective sleep quality, time to fall asleep, sleep time, sleep efficiency, sleep disorders, hypnotic drugs, and daytime function. The higher the total score, the worse the sleep quality.
Resilience | 2023.6.1-2024.7.1
  The Corner Davidson Resilience Scale (CDRISC) consists of 10 items and uses the Likert 5-point scoring system. A score of 0-4 indicates "never", "rarely", "sometimes", "often", and "always", with higher scores indicating higher levels of psychological resilience.

CONTACTS AND LOCATIONS:
Overall Officials: DanTing Chen, Principal Investigator — Fujian Medical University
Locations (1):
- Fujian provincial hospital, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No